CLINICAL TRIAL: NCT03288675
Title: The Effects of Accelerated Intermittent Thetaburst Stimulation Followed by a Cognitive Control Training in Treatment Resistant Unipolar Depressed Patients
Brief Title: Stepped Care AiTBS 2 Depression Study (Ghent)
Acronym: aiTBS2-Ghent
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Ghent (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Triple | Purpose: Treatment
Other Study IDs: BC-1812
Record Dates: First submitted 2017-07-14; First posted 2017-09-20 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Depressive Disorder, Major; Treatment Resistant Depression; Melancholia
Keywords: Major depressive disorder; Treatment resistant depression; Accelerated intermittent thetaburst stimulation; Cognitive control training; Neuroimaging
MeSH Terms: conditions — Depressive Disorder, Major; Depressive Disorder, Treatment-Resistant; Depressive Disorder | interventions — Selective Serotonin Reuptake Inhibitors

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Active aiTBS - active CCT+SSRI (Active Comparator): Patients receive active aiTBS treatment in the first week, and starting from week 3 receive active CCT for a period of 4 weeks in combination with an antidepressant (SSRI)
  Interventions: Device: aiTBS; Behavioral: CCT; Drug: SSRI
- Active aiTBS - sham CCT+SSRI (Experimental): Patients receive active aiTBS treatment in the first week, and starting from week 3 receive a control training for a period of 4 weeks in combination with an antidepressant (SSRI)
  Interventions: Device: aiTBS; Drug: SSRI
- Sham aiTBS - aiTBS - active CCT+SSRI (Experimental): Patients receive sham aiTBS treatment in the first week, real aiTBS treatment in the third week, and starting from the fifth week receive CCT for a period of 4 weeks in combination with an antidepressant (SSRI)
  Interventions: Device: aiTBS; Behavioral: CCT; Drug: SSRI
- Sham aiTBS - aiTBS - sham CCT+SSRI (Experimental): Patients receive sham aiTBS treatment in the first week, real aiTBS treatment in the third week, and starting from the fifth week control training for a period of 4 weeks in combination with an antidepressant (SSRI)
  Interventions: Device: aiTBS; Drug: SSRI

INTERVENTIONS:
Device: aiTBS — In the active aiTBS arm, the patients will receive 100 cycli of thetaburst trains of 2s, separated by an inter-train-interval of 6 seconds, delivered on the left dorsolateral prefrontal cortex (DLPFC; i.e. 3000 pulses per session). On each stimulation day, a given patient will receive 5 sessions with a between-session interval of 15 minutes. The treatment protocol of in total 20 aiTBS sessions will be spread over 4 days (i.e. 60.000 pulses in total). The sham coil has been specifically developed to mimic the real one.
  Other Names: accelerated intermittent thetaburst stimulation
Behavioral: CCT — By training working memory processing, the CCT aims at modulating similar prefrontal cortex regions as being stimulated previously by aiTBS, namely the DLPFC. thereby possibly stabilizing clinical effects of aiTBS over time. In total 20 sessions of CCT vs. control training (of approximately 25 minutes per session), will be spread over a period of 4 weeks.
  Other Names: cognitive control training
  Arms: Active aiTBS - active CCT+SSRI; Sham aiTBS - aiTBS - active CCT+SSRI
Drug: SSRI — All patients will be prescribed antidepressant medication (SSRI) again when starting the CCT (vs. control training).
  Other Names: selective serotonin reuptake inhibitor

SUMMARY:
Antidepressant-free unipolar melancholic depressed patients (at least stage 2 treatment-resistant) will be selected by a certified psychiatrist, who will administer (semi-)structured clinical interviews. Because concomitant antidepressant treatment can confound outcome results, all patients will go through a medication washout before entering the study and they will be free from any antidepressant, neuroleptic and mood stabilizer for at least two weeks before entering the treatment protocol. Only habitual benzodiazepine agents will be allowed.

STEP 1: Patients will be treated with in total 20 accelerated intermittent Theta Burst Stimulation (aiTBS) sessions (3000 pulses/session) over the left dorsolateral prefrontal cortex, which will be spread over 4 days. On each stimulation day, a given patient will receive 5 sessions with a between-session delay of 15 minutes. Patients will be randomized to receive either the real aiTBS or sham treatment (first week). However, the sham group will receive real aiTBS treatment with 10 days' time interval. The investigators expect that real aiTBS treatment and not sham will result in a significant and clinical meaningful response.

STEP 2: To optimize treatment and reduce relapse following the iTBS treatment, in a stepped care approach, all patients then continue with cognitive control training (CCT) ten days later. This CCT consists of 20 sessions, spread over 4 weeks. Patients will be randomized to receive either real CCT or a control training. During this follow-up treatment, all patients will be prescribed antidepressant medication (SSRI) again. As iTBS treatment effects are known to decline over time, the investigators expect that combining aiTBS with a follow-up CCT therapy will stabilize the clinical effects over time compared to receiving the iTBS treatment alone.

For baseline comparisons, patients will be closely matched for gender and age with never-depressed, medication-free healthy volunteers. No volunteer will undergo treatment.

ELIGIBILITY:
Inclusion Criteria:

* Antidepressant-free unipolar major depression with melancholic features
* Not responding to at least two trials with an antidepressant
* Aged between 18-65 years old

Exclusion Criteria:

* Depression with bipolar/psychotic features
* Dysthymia
* Severe personality disorders
* Active substance abuse/dependence within a year prior to inclusion
* Pregnancy or without effective anticonception for the duration of the trial
* ECT non-responder
* No response to more than 9 antidepressants
* Any neurological condition
* Any implanted electronic device susceptible for magnetic field radiation (e.g. pacemaker)
* Any implanted metal device in the head region
* Current or past history of epilepsy
* Neurosurgical interventions
* Known allergic reaction to radiotracers or associated compounds

Healthy volunteers may be accepted as control subjects.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 68 (Actual)
Dates: Start 2017-10-05 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
Changes in depression severity - clinician-rated | Intake, baseline (D0), 3 days after aiTBS or sham (+/-D7), 10 days after aiTBS or sham (+/-D14), [for the sham group 3 days (+/-D21) and 10 days after active aiTBS (+/-D28)], after CCT (+/-D42; for the sham group +/-D56), 3 & 6 months follow-up
  17-item Hamilton Rating Scale for Depression (HRSD)

SECONDARY OUTCOMES:
Changes in depression severity - self-report | Intake, baseline (D0), 3 days after aiTBS or sham (+/-D7), 10 days after aiTBS or sham (+/-D14), [for the sham group 3 days (+/-D21) and 10 days after active aiTBS (+/-D28)], after CCT (+/-D42; for the sham group +/-D56), 3 & 6 months follow-up
  Beck Depression Inventory (BDI-II)
Changes in suicidal thoughts - clinician-rated | Intake, baseline (D0), 3 days after aiTBS or sham (+/-D7), 10 days after aiTBS or sham (+/-D14), [for the sham group 3 days (+/-D21) and 10 days after active aiTBS (+/-D28)], after CCT (+/-D42; for the sham group +/-D56), 3 & 6 months follow-up
  Scale for suicidal ideation (SSI)
Changes in melancholic features - clinician-rated | Intake, baseline (D0), 3 days after aiTBS or sham (+/-D7), 10 days after aiTBS or sham (+/-D14), [for the sham group 3 days (+/-D21) and 10 days after active aiTBS (+/-D28)], after CCT (+/-D42; for the sham group +/-D56), 3 & 6 months follow-up
  Clinical outcomes in routine evaluation (CORE)
Changes in hopelessness - self-report | Baseline (D0), 3 days after aiTBS or sham (+/-D7), 10 days after aiTBS or sham (+/-D14), [for the sham group 3 days (+/-D21) and 10 days after active aiTBS (+/-D28)], after CCT (+/-D42; for the sham group +/-D56), 3 & 6 months follow-up
  Beck hopelessness scale (BHS)
Changes in anxiety features - self-report | Baseline (D0), 3 days after aiTBS or sham (+/-D7), 10 days after aiTBS or sham (+/-D14), [for the sham group 3 days (+/-D21) and 10 days after active aiTBS (+/-D28)], after CCT (+/-D42; for the sham group +/-D56), 3 & 6 months follow-up
  State/Trait Anxiety Inventory (STAI)
Changes in remission from depression - self-report | Baseline (D0), 3 days after aiTBS or sham (+/-D7), 10 days after aiTBS or sham (+/-D14), [for the sham group 3 days (+/-D21) and 10 days after active aiTBS (+/-D28)], after CCT (+/-D42; for the sham group +/-D56), 3 & 6 months follow-up
  Remission from Depression Questionnaire (RDQ)
Changes in ruminative thinking (trait) - self-report | Baseline (D0), 10 days after aiTBS or sham (+/-D14), [for the sham group 10 days after active aiTBS (+/-D28)], after CCT (+/-D42; for the sham group +/-D56), 3 & 6 months follow-up
  Ruminative Responses Scale (RRS)
Changes in hedonia - self-report | Baseline (D0), 10 days after aiTBS or sham (+/-D14), [for the sham group 10 days after active aiTBS (+/-D28)], after CCT (+/-D42; for the sham group +/-D56), 3 & 6 months follow-up
  Temporal Experience of Pleasure Scale (TEPS)
Changes in anhedonia - self-report | Baseline (D0), 10 days after aiTBS or sham (+/-D14), [for the sham group 10 days after active aiTBS (+/-D28)], after CCT (+/-D42; for the sham group +/-D56), 3 & 6 months follow-up
  Snaith-Hamilton Pleasure Scale (SHAPS)
Changes in perceived stress - self-report | Baseline (D0), 10 days after aiTBS or sham (+/-D14), [for the sham group 10 days after active aiTBS (+/-D28)], after CCT (+/-D42; for the sham group +/-D56), 3 & 6 months follow-up
  Perceived Stress Scale (PSS)
Changes in responses to positive affect - self-report | Baseline (D0), 10 days after aiTBS or sham (+/-D14), [for the sham group 10 days after active aiTBS (+/-D28)], after CCT (+/-D42; for the sham group +/-D56), 3 & 6 months follow-up
  Responses to Positive Affect Scale (RPA)
Changes in cognitive emotion regulation - self-report | Baseline (D0), 10 days after aiTBS or sham (+/-D14), [for the sham group 10 days after active aiTBS (+/-D28)], after CCT (+/-D42; for the sham group +/-D56), 3 & 6 months follow-up
  Cognitive Emotion Regulation Questionnaire (CERQ)
Changes in temperament and character - self-report | Intake, 10 days after aiTBS or sham (+/-D14)
  Temperament and Character Inventory (TCI)
Differences in adverse effects following aiTBS vs. sham - self-report | 10 days after aiTBS or sham (+/-D14), [for the sham group 10 days after active aiTBS (+/-D28)]
  Adverse effects questionnaire
Changes in regional grey matter volume using structural MRI | Baseline (D0), 10 days after aiTBS or sham (+/-D14)
  The analysis will be done using voxel-based morphometry
Changes in regional white matter microstructure and structural connectivity | Baseline (D0), 10 days after aiTBS or sham (+/-D14)
  The analysis will be done using diffusion tensor imaging (DTI)
Neuronal safety/ changes in neurometabolite concentrations in left-prefrontal tissues using MRS | Baseline (D0), 10 days after aiTBS or sham (+/-D14)
  The analysis will be evaluated using 1H MR spectroscopy
Changes in functional activity connectivity at rest and during tasks in which self-referential social evaluations are presented via headphones in the scanner | Baseline (D0), 10 days after aiTBS or sham (+/-D14)
  The analysis will be evaluated using resting state and task fMRI
Changes in state-dependent ruminative thinking due to hearing self-referential social evaluations presented via headphones in the scanner - self-report | Baseline (D0), 10 days after aiTBS or sham (+/-D14)
  Before entering the scanner, and following each resting state fMRI (i.e. before hearing self-referential social evaluations and after hearing these evaluations), perseverative thinking will be assessed using the perseverative thinking questionnaire (PTQ).
Changes in state-dependent mood due to hearing self-referential social evaluations presented via headphones in the scanner - self-report | Baseline (D0), 10 days after aiTBS or sham (+/-D14)
  Before entering the scanner, and following each resting state fMRI (i.e. before hearing self-referential social evaluations and after hearing these evaluations), mood will be assessed using visual analogue scales (VAS).
Changes in the regional 5-HT transporter system | Baseline (D0), 3 days after aiTBS or sham (+/-D7), 10 days after aiTBS or sham (+/-D14)
  C11 DASB PET
Changes in reward processing as measured with EEG /ERP | Baseline (D0), 10 days after active aiTBS in both groups (+/-D14 for the active group, +/-D28 for the sham group)
  128 channel EEG during doors gambling task to assess effects on reward processing.
Evaluation of cognitive side-effects following iTBS vs. sham using the CANTAB battery | Baseline (D0), 3 days after aiTBS or sham (+/-D7)
  CANTAB battery administration (i.e. motor screening, delayed matching to sample, rapid visual information processing, one touch stockings of Cambridge, spatial working memory).
Changes in reward processing - behavioral assessment | Baseline (D0), 10 days after aiTBS or sham (+/-D14), [for the sham group 10 days after active aiTBS (+/-D28)], after CCT (+/-D42; for the sham group +/-D56)
  Cambridge Gambling Task (CGT; CANTAB battery)
Changes in working memory - behavioral assessment of near transfer | Baseline (D0), 10 days after active aiTBS in both groups (+/-D14 for the active group, +/-D28 for the sham group), after CCT (+/-D42; for the sham group +/-D56)
  Non-adaptive PASAT (naPASAT)
Changes in state-dependent mood - self-report following naPASAT | Baseline (D0), 10 days after active aiTBS in both groups (+/-D14 for the active group, +/-D28 for the sham group), after CCT (+/-D42; for the sham group +/-D56)
  Visual analogue scales (VAS) administered following completion of the naPASAT
Changes in spatial working memory - behavioral assessment of far transfer | Baseline (D0), 10 days after active aiTBS in both groups (+/-D14 for the active group, +/-D28 for the sham group), after CCT (+/-D42; for the sham group +/-D56)
  Spatial working memory (SWT; CANTAB battery)
Changes in state-dependent mood during CCT vs. control training | Following each of the 20 CCT or control trainings (spread over +/- D15 up to D42 for the active group; spread over +/- D29 up to D56 for the sham group)
  Visual analogue scales (VAS) administered following completion of the CCT (or control training)
Predictive influence of single nucleotide polymorphisms on treatment outcome - genetics using a saliva sample | At baseline (D0)
  SNP analysis
Predictive influence of treatment expectancy on treatment response - self-report | After the first aiTBS or sham session (D1), after the first CCT or control session (+/- D15 for the active group, +/-D29 for the sham group)
  Credibility and Expectancy Questionnaire (CEQ)

CONTACTS AND LOCATIONS:
Overall Officials: Chris Baeken, Prof., Principal Investigator — Ghent University, University Hospital Ghent; Ernst Koster, Prof., Principal Investigator — University Ghent; Rudi De Raedt, Prof., Principal Investigator — University Ghent; Gilles Pourtois, Prof., Principal Investigator — University Ghent; Marie-Anne Vanderhasselt, Prof., Principal Investigator — Ghent University, University Hospital Ghent
Locations (1):
- University Hospital Ghent, Ghent, East-Flanders, Belgium

IPD SHARING:
Plan to Share IPD: No